CLINICAL TRIAL: NCT00824330
Title: The Use of a Home-based Walking Program to Treat Orthostatic Hypotension in Older Adults With Type 2 Diabetes
Brief Title: Home-Based Walking Study in Older Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kenneth Madden, Head, VGH Division of Geriatric Medicine, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H08-02237
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular; Diabetes; Orthostatic Hypotension; Type 2 Diabetes
Keywords: Aging; Type 2 diabetes; exercise; walking; glucose metabolism; arterial baroreceptors; heart rate variability; cerebral autoregulation; tilt table study; transcranial Doppler; autonomic nervous system
MeSH Terms: conditions — Diabetes Mellitus; Hypotension, Orthostatic; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control Phase; Exercise Phase (Other): Participants act as their own control.
  Control Phase:
  Participants will not change their activity during the 3 month control phase (defined as no strength training and less than 30 minutes brisk walking/moderate exercise per week, no vigorous exercise) Baseline measures will be obtained.
  Exercise Phase:
  This phase will consist of a Titration phase followed by an Intervention Phase. During the Titration phase, under the guidance of a trainer, subjects will increase their number of steps by 20% per week until they have reached 10,000 steps or 3 months have passed. During the Intervention Phase subjects will continue to walk 10,000 steps (or the number of steps they reached in the Titration phase).
  Interventions: Behavioral: Control Phase; Exercise Phase

INTERVENTIONS:
Behavioral: Control Phase; Exercise Phase — After the completion of the control phase and at the start of the titration phase of the study, participants will be given pedometers and log books, then contacted on a regular basis to help insure compliance with the goal of walking 10,000 steps per day.

SUMMARY:
Older persons with diabetes have a harder time maintaining blood pressure when standing up. When blood pressure drops when standing up, fainting may occur. This study will see how regular exercise can improve the ability of the body to keep blood pressure up when standing. We want to see how this improvement varies with a home-based walking program.

DETAILED DESCRIPTION:
Detailed Summary

1. PURPOSE: Older adults with diabetes faint frequently, due to an impairment in the cardiovascular control mechanisms (arterial baroreceptor function, autonomic nervous system function and cerebral autoregulation) that prevent syncope. The purpose of this study is to examine the ability of a home based walking program to reverse these impairments.
2. HYPOTHESES: a) A home-based walking program will improve the compensatory cardiovascular responses that prevent syncope in older adults with Type 2 diabetes. A moderate, regular exercise program will:

   * increase arterial baroreflex sensitivity
   * increase heart rate variability (marker of autonomic nervous system function)
   * decrease cerebrovascular resistance
   * improve cerebral autoregulation during upright tilt. b) There will be relationship between the improvement in compensatory cardiovascular responses and regular exercise.

     c) Design of more practicable training prescriptions than that used in a research setting.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 5 years treated with diet alone or oral agents
* Nonsmoker for at least 5 years
* Subjects must be sedentary (as defined by no strength training and less than 30 minutes brisk walking/moderate exercise per week and no vigorous exercise in the preceding 6 months)
* All subjects will have a fasting glucose of <12 mM and a hemoglobin A1c < 8.5%
* Orthostatic hypotension defined as a decrease in systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of at least 10 mm Hg within 3 minutes of assuming an upright posture on the initial screening visit as per current American Academy of Neurology guidelines.

Exclusion Criteria:

* Abnormalities on complete blood count, electrolytes or creatinine, on resting ECG, treadmill exercise stress test
* Significant pulmonary, exercise-limiting orthopedic or neurological impairment
* Evidence of valvular disease, exercise-induced syncope, angina, arrhythmias or peripheral vascular disease
* Poor blood pressure control as defined as systolic blood pressure greater than or equal to 160 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg
* Total cholesterol/HDL cholesterol greater than or equal to 5.0 or LDL cholesterol greater than or equal to 4.21 mmol/L
* Peripheral neuropathy severe enough to cause discomfort (for safety reasons)
* Overt diabetic nephropathy excluding subjects with a urine albumin to creatinine ratio of greater than 2.0 in men or 2.8 in women
* Diabetic retinopathy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity (central and peripheral) | Measured at Baseline, 3 months after control phase and after 3 months of Intervention phase
Drop in middle cerebral artery velocity with upright tilting | Measured at Baseline, 3 months after control phase and after 3 months of Intervention phase
Drop in blood pressure with upright tilt | Measured at Baseline, 3 months after control phase and after 3 months of Intervention phase
Arterial baroreflex sensitivity | Measured at Baseline, 3 months after control phase and after 3 months of Intervention phase

SECONDARY OUTCOMES:
Fasting blood glucose, HgbA1C | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
VO2max | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
Dynamometry measures of muscle strength | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
Resting and maximal heart rate | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
Waist to hip ratio, BMI | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
Lean body mass/% fat | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
Catecholamines | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.
Increase in Gosling's pulsatility index | Measured at Baseline, 3 month after control phase and after 3 months of Intervention phase.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Madden, Principal Investigator — University of British Columbia; Karim Miran-Khan, Study Director — University of British Columbia; Janet McElhaney, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - VITALiTY Research Centre - VGH Research Pavilion, Vancouver, British Columbia
  - Dr. Scott Lear's Lab, Simon Fraser University, Harbour, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No